CLINICAL TRIAL: NCT05368311
Title: Effect of a Protein Intake on Weight Loss of Overweight/Obese Adults
Acronym: COLABOCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLABOCO
Record Dates: First submitted 2022-03-03; First posted 2022-05-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2021-12

CONDITIONS: Obesity; Weight Loss; Protein
Keywords: Protein; Weight loss; Obesity; Overweight; Satiety
MeSH Terms: conditions — Obesity; Weight Loss; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving dietary recommendations including protein enriched bars . (Experimental): Experimental group will consume two protein enriched bars per day during 12 weeks. First bar will be consumed 45 minutes before lunch and second bar will be consumed 45 minutes before dinner.
  Interventions: Other: Dietary recommendations including protein enriched bars
- Group receiving dietary recommendations without protein enriched bars. (Placebo Comparator): Placebo group will follow just dietary recommendations during 12 weeks.
  Interventions: Other: Dietary recommendations without protein enriched bars

INTERVENTIONS:
Other: Dietary recommendations including protein enriched bars — Volunteers allocated in the experimental group will receive dietary recommendations and 2 protein enriched bars per day to be eaten 45 minutes before lunch and dinner.
  Arms: Group receiving dietary recommendations including protein enriched bars .
Other: Dietary recommendations without protein enriched bars — Volunteers allocated in the experimental group will receive dietary recommendations.
  Arms: Group receiving dietary recommendations without protein enriched bars.

SUMMARY:
Obesity is considered the epidemic of the 21st century. Obesity is a multifactorial disease and the most important risk factors are poor diet and sedentary lifestyle. An excessive body weight contributes to increase the risk of suffering from other diseases and mortality rates. Therefore, the prevention and control of excessive body weight as well as its comorbidities are essential. In this sense, the principal strategy to treat obesity is to improve dietary habits and increase physical activity. However, the rate of obesity continues rising. In order to deal with this problem, new strategies to combat obesity are being investigated, such as the investigation of new bioactive compounds with satiating capacity that can be included in healthy dietary patterns to improve adherence to dietary treatments.

Considering this background, the main objective of this research is to assess the effect of daily consumption of protein rich bars accompanied by healthy dietary recommendations on weight loss of overweight/obese adult men and women.

DETAILED DESCRIPTION:
This study is designed as a 12-week, randomised, parallel study, focused on overweight/obese men and women between 20 and 65 years old.

All participants attend the Nutrition Intervention Unit of the Center for Nutrition Research in the University of Navarra for the screening visit and 4 more times during the intervention (week 1, 4, 8 and 12 of study).

Screening visit: evaluation of the inclusion criteria. Volunteers who meet the inclusion criteria are provided with a feces collection kit, urine collection kit, food frequency questionnaire, visual analogue scale and minnesota physical activity questionnaire. Moreover, they are randomly assigned to one of the two intervention groups:

* Control group: healthy dietary recommendations.
* Experimental group: healthy dietary recommendations + 2 protein rich bars/day

Clinical investigation day 1 (week 1): The volunteer attend the Nutrition Intervention Unit in fasting condition. Each volunteer is asked to provide the fece and urine samples, and completed questionnaires provided in screening visit. Then, anthropometric, body composition, densitometry and blood pressure measurements are taken and the gastrointestinal symptoms questionnaire is completed. After that, volunteer is provided with healthy dietary recommendations only or dietary recommendations and protein rich bars, depending on the allocated intervention group. Moreover, volunteer is provided with visual analogue scale to be completed for the Clinical investigation day 2.

Clinical investigation day 2 (week 4): The volunteer attend the Nutrition Intervention Unit. The volunteer is asked to provide the visual analogue scale. Then, gastrointestinal symptoms questionnaire is completed and the adherence to the study is assessed. Then, body weight and blood pressure are measured. Volunteer is provided with fece and urine collection kits, food frequency questionnaire, minnesota physical activity questionnaire and visual analogue scale, to be completed for the Clinical investigation day 3. Finally, volunteers allocated in experimental group are provided with protein rich bars.

Clinical investigation day 3 (week 8): The volunteer attend the Nutrition Intervention Unit in fasting condition. Each volunteer is asked to provide the fece and urine samples, and completed questionnaires provided in Clinical investigation day 2. After that, the adherence to the study is assessed. Then, anthropometric, body composition, densitometry and blood pressure measurements are taken and the gastrointestinal symptoms questionnaire is completed. Volunteer is provided with fece and urine collection kits, as well as food frequency questionnaire, minnesota physical activity questionnaire and visual analogue scale to be completed for the Clinical investigation day 4. Finally, volunteers allocated in experimental group are provided with protein rich bars.

Clinical investigation day 4 (week 12): The volunteer attend the Nutrition Intervention Unit in fasting condition. Each volunteer is asked to provide the fece and urine samples, and completed questionnaires provided in Clinical investigation day 3. After that, the adherence to the study is assessed. Then, anthropometric, body composition, densitometry and blood pressure measurements are taken and the gastrointestinal symptoms questionnaire is completed.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with BMI between 24.9 and 34.9 kg/m2.
* Physical examination and vital signs normal or clinically irrelevant to the study.
* Volunteers undergoing pharmacological treatment will be included if the dose is stable for at least 3 months before the start of the study, excluding treatments that alter gastrointestinal function and antidiabetics.
* Subjects must be able to understand and be willing to sign the informed consent, as well as comply with all the procedures and requirements of the study.
* Present a stable weight (+/-3kg) in the last three months before the start of the study.

Exclusion Criteria:

* Subjects with relevant functional or structural abnormalities of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory or malabsorption diseases, hiatal hernia, reflux, etc.
* Subjects with a high alcohol intake, more than 14 units (women) and 20 units (men).
* Women who are breastfeeding or pregnant.
* Subjects who have undergone surgical interventions with permanent sequelae in the digestive system (for example, gastroduodenostomy).
* Subjects with liver disease.
* Subjects with some type of cancer or undergoing treatment for it, or who have not had a period of at least 5 years since its eradication.
* Subjects with allergies to any component of the product under study or any other food that interferes and makes it difficult to monitor the study.
* Subjects who present some type of cognitive and/or psychic impairment.
* Subjects in whom poor collaboration is expected or who, in the opinion of the investigator, have difficulties in following the study procedures.
* Subjects who work night shifts.
* Subjects who follow some type of supplementation that interferes with the study.
* Subjects who are immersed in some treatment for weight loss.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Balanced in men and women.
Enrollment: 64 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change of weight from baseline to week 4 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Weight of participants in fasting condition will be analyzed by bioimpedance and reported in kg.
Change of weight from baseline to week 8 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Weight of participants in fasting condition will be analyzed by bioimpedance and reported in kg.
Change of weight from baseline to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Weight of participants in fasting condition will be analyzed by bioimpedance and reported in kg.
Change of weight from week 4 to week 8 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 2 (after 4 week of intervention) compared to Clinical Investigation Day 3(after 8 weeks of intervention).
  Weight of participants in fasting condition will be analyzed by bioimpedance and reported in kg.
Change of weight from week 4 to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 2 (after 4 week of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Weight of participants in fasting condition will be analyzed by bioimpedance and reported in kg.
Change of weight from week 8 to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 week of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Weight of participants in fasting condition will be analyzed by bioimpedance and reported in kg.

SECONDARY OUTCOMES:
Change of body fat percentage from baseline to week 8 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Body fat of participants in fasting condition will be analyzed by bioimpedance and reported in percentage.
Change of body fat percentage from baseline to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Body fat of participants in fasting condition will be analyzed by bioimpedance and reported in percentage.
Change of body fat percentage from week 8 to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Body fat of participants in fasting condition will be analyzed by bioimpedance and reported in percentage.
Change of body fat kilograms from baseline to week 8 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Body fat of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body fat kilograms from baseline to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Body fat of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body fat kilograms from week 8 to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Body fat of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body muscle mass from baseline to week 8 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Muscle mass of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body muscle mass from baseline to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Muscle mass of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body muscle mass from week 8 to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Muscle mass of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body lean mass from baseline to week 8 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Lean mass of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body lean mass from baseline to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Lean mass of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body lean mass from week 8 to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Lean mass of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body water mass from baseline to week 8 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Body water of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body water mass from baseline to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Body water of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body water mass from week 8 to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Body water of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of body water percentage from baseline to week 8 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Body water of participants in fasting condition will be analyzed by bioimpedance and reported in percentage.
Change of body water percentage from baseline to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Body water of participants in fasting condition will be analyzed by bioimpedance and reported in percentage.
Change of body water percentage from week 8 to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Body water of participants in fasting condition will be analyzed by bioimpedance and reported in percentage.
Change of bone mass from baseline to week 8 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Bone mass of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of bone mass from baseline to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Bone mass of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Change of bone mass from week 8 to week 12 (bioimpedance) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Bone mass of participants in fasting condition will be analyzed by bioimpedance and reported in kilograms.
Height at baseline | The Time Frame contains one time point: screening visit.
  Height of participants will be measured by stadiometer and reported in meters.
Change of waist circumference from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Waist circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change of waist circumference from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Waist circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change of waist circumference from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Waist circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change of hip circumference from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Hip circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change of hip circumference from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Hip circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change of hip circumference from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Hip circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change of neck circumference from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Neck circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change of neck circumference from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Neck circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change of neck circumference from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Neck circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Change of systolic blood pressure from baseline to week 4 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Systolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change of systolic blood pressure from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Systolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change of systolic blood pressure from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Systolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change of systolic blood pressure from week 4 to week 8 | The Time Frame contains two time points: Clinical Investigation Day 2 (after 4 weeks of intervention) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Systolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change of systolic blood pressure from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Systolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change of diastolic blood pressure from baseline to week 4 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Diastolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change of diastolic blood pressure from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Diastolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change of diastolic blood pressure from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Diastolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change of diastolic blood pressure from week 4 to week 8 | The Time Frame contains two time points: Clinical Investigation Day 2 (after 4 weeks of intervention) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Diastolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change of diastolic blood pressure from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Diastolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Change of heart rate from baseline to week 4 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Heart rate of participants in fasting condition will be analyzed by electronic tensiometer and reported in beats per minute.
Change of heart rate from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Heart rate of participants in fasting condition will be analyzed by electronic tensiometer and reported in beats per minute.
Change of heart rate from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Heart rate of participants in fasting condition will be analyzed by electronic tensiometer and reported in beats per minute.
Change of heart rate from week 4 to week 8 | The Time Frame contains two time points: Clinical Investigation Day 2 (after 4 weeks of intervention) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Heart rate of participants in fasting condition will be analyzed by electronic tensiometer and reported in beats per minute.
Change of heart rate from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Heart rate of participants in fasting condition will be analyzed by electronic tensiometer and reported in beats per minute.
Change of body fat mass in percentage from baseline to week 8 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of body fat mass of participants in fasting condition will be analyzed by densitometry machine and reported in percentage.
Change of body fat mass in percentage from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of body fat mass of participants in fasting condition will be analyzed by densitometry machine and reported in percentage.
Change of body fat mass in percentage from week 8 to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of body fat mass of participants in fasting condition will be analyzed by densitometry machine and reported in percentage.
Change of body fat mass in kg from baseline to week 8 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of body fat mass of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of body fat mass in kg from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of body fat mass of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of body fat mass in kg from week 8 to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of body fat mass of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of lean mass in kg from baseline to week 8 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of body fat mass of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of lean mass in kg from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of body fat mass of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of lean mass in kg from week 8 to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of body fat mass of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of lean mass in kg from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of lean mass of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of bone mineral concentration from baseline to week 8 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of bone mineral concentration of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of bone mineral concentration from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bone mineral concentration of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of bone mineral concentration from week 8 to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bone mineral concentration of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of bone mineral density from baseline to week 8 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of bone mineral density of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of bone mineral density from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bone mineral density of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of bone mineral density from week 8 to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bone mineral density of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of visceral mass from baseline to week 8 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of visceral mass of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of visceral mass from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of visceral mass density of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of visceral mass from week 8 to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of visceral mass of participants in fasting condition will be analyzed by densitometry machine and reported in kilograms.
Change of L1-L4 bone mineral density from baseline to week 8 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of L1-L4 bone mineral density of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of L1-L4 bone mineral density from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of L1-L4 bone mineral density of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of L1-L4 bone mineral density from week 8 to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of L1-L4 bone mineral density of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of total bone mineral density of femur from baseline to week 8 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of bone mineral density of femur of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of total bone mineral density of femur from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bone mineral density of femur of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of total bone mineral density of femur from week 8 to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bone mineral density of femur of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of bone mineral density of femur neck from baseline to week 8 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of bone mineral density of femur neck of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of bone mineral density of femur neck from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bone mineral density of femur neck of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of bone mineral density of femur neck from week 8 to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bone mineral density of femur neck of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of bone mineral density of radius from baseline to week 8 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of bone mineral density of radius of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of bone mineral density of radius from baseline to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bone mineral density of radius of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of bone mineral density of radius from week 8 to week 12 (densitometry) | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bone mineral density of radius of participants in fasting condition will be analyzed by densitometry machine and reported in g/m2.
Change of glucose concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of glucose levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of glucose concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of glucose levels of participants in fasting condition will be analyzed by absorptiometry and reported in mg/dL.
Change of glucose concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of glucose levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of total cholesterol concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of total cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of total cholesterol concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of total cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of total cholesterol concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of total cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of HDL cholesterol concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of HDL cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of HDL cholesterol concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of HDL cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of HDL cholesterol concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of HDL cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of LDL cholesterol concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of LDL cholesterol levels of participants in fasting condition will be analyzed by Friedewald formula and reported in mg/dL.
Change of LDL cholesterol concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of LDL cholesterol levels of participants in fasting condition will be analyzed by Friedewald formula and reported in mg/dL.
Change of LDL cholesterol concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of LDL cholesterol levels of participants in fasting condition will be analyzed by Friedewald formula and reported in mg/dL.
Change of triglyceride concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of triglyceride levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of triglyceride concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of triglyceride levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of triglyceride concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of triglyceride levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of alanine aminotransferase concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of alanine aminotransferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in U/L.
Change of alanine aminotransferase concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of alanine aminotransferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in U/L.
Change of alanine aminotransferase concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of alanine aminotransferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in U/L.
Change of aspartate aminotransferase concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of aspartate aminotransferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Change of aspartate aminotransferase concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of aspartate aminotransferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in U/L.
Change of aspartate aminotransferase concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of aspartate aminotransferase levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in U/L.
Change of homocysteine concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of homocysteine levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in μmol/L.
Change of homocysteine concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of homocysteine levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in μmol/L..
Change of homocysteine concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of homocysteine levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in μmol/L..
Change of C-reactive protein concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of C-reactive protein levels of participants in fasting condition will be analyzed by ELISA and reported in mg/L.
Change of C-reactive protein concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of C-reactive protein levels of participants in fasting condition will be analyzed by ELISA and reported in mg/L.
Change of C-reactive protein concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of C-reactive protein levels of participants in fasting condition will be analyzed by ELISA and reported in mg/L.
Change of hemogram concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of hemogram levels of participants in fasting condition will be analyzed by biochemical autoanalyzer.
Change of hemogram concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of hemogram levels of participants in fasting condition will be analyzed by biochemical autoanalyzer.
Change of hemogram concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of hemogram levels of participants in fasting condition will be analyzed by biochemical autoanalyzer.
Change of albumin concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of albumin levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer.
Change of albumin concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of albumin levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer.
Change of albumin concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of albumin levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer.
Change of creatinine concentration from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 8 weeks of intervention).
  Change of creatinine levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer and reported in μmol/L.
Change of creatinine concentration from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of creatinine levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer and reported in μmol/L.
Change of creatinine concentration from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of creatinine levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer and reported in μmol/L.
Change of physical activity level from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of physical activity level of participants will be analyzed by Minnesota physical activity questionnaire and reported in mets.
Change of physical activity level from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of physical activity level of participants will be analyzed by Minnesota physical activity questionnaire and reported in mets.
Change of physical activity level from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of physical activity level of participants will be analyzed by Minnesota physical activity questionnaire and reported in mets.
Change of dietary intake from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of dietary intake of participants will be analyzed by Food Frequency Questionnaire.
Change of dietary intake from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of dietary intake of participants will be analyzed by Food Frequency Questionnaire.
Change of dietary intake from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of dietary intake of participants will be analyzed by Food Frequency Questionnaire.
Change of hunger from baseline to week 4 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  The change in hunger of participants will be analyzed by Hunger-Satiety Visual Analogue Scale (VAS). The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in hunger scale means better outcome.
Change of hunger from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in hunger of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in hunger scale means better outcome.
Change of hunger from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in hunger of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in hunger scale means better outcome.
Change of hunger from week 4 to week 8 | The Time Frame contains two time points: Clinical Investigation day 2 (after 4 weeks of intervention) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in hunger of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in hunger scale means better outcome.
Change of hunger from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in hunger of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in hunger scale means better outcome.
Change of fullness from baseline to week 4 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  The change in fullness of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in fullness scale means better outcome.
Change of fullness from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in fullness of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in fullness scale means better outcome.
Change of fullness from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in fullness of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in fullness scale means better outcome.
Change of fullness from week 4 to week 8 | The Time Frame contains two time points: Clinical Investigation day 2 (after 4 weeks of intervention) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in fullness of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in fullness scale means better outcome.
Change of fullness from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in fullness of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in fullness scale means better outcome.
Change of satisfaction sensation from baseline to week 4 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  The change in satisfaction sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in satisfaction scale means better outcome.
Change of satisfaction sensation from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in satisfaction sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in satisfaction scale means better outcome.
Change of satisfaction sensation from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in satisfaction sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in satisfaction scale means better outcome.
Change of satisfaction sensation from week 4 to week 8 | The Time Frame contains two time points: Clinical Investigation day 2 (after 4 weeks of intervention) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in satisfaction sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in satisfaction scale means better outcome.
Change of satisfaction sensation from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in satisfaction sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in satisfaction scale means better outcome.
Change of want to eat something else sensation from baseline to week 4 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  The change in want to eat something else sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in want to eat something else scale means better outcome.
Change of want to eat something else sensation from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in want to eat something else sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in want to eat something else scale means better outcome.
Change of want to eat something else sensation from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in want to eat something else sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in want to eat something else scale means better outcome.
Change of want to eat something else sensation from week 4 to week 8 | The Time Frame contains two time points: Clinical Investigation day 2 (after 4 weeks of intervention) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in want to eat something else sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in want to eat something else scale means better outcome.
Change of want to eat something else sensation from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in want to eat something else sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in want to eat something else scale means better outcome.
Change of thirst sensation from baseline to week 4 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  The change in thirst sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in want to eat something else scale means better outcome.
Change of thirst sensation from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in thirst sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm.
Change of thirst sensation from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in thirst sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm.
Change of thirst sensation from week 4 to week 8 | The Time Frame contains two time points: Clinical Investigation day 2 (after 4 weeks of intervention) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in thirst sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm.
Change of thirst sensation from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in thirst sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm.
Change of gastrointestinal symptoms from baseline to week 4 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  The change in gastrointestinal symptoms of participants will be analyzed by gastrointestinal symptoms questionnaire. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in the gastrointestinal symptoms means better outcome.
Change of gastrointestinal symptoms from baseline to week 8 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in gastrointestinal symptoms of participants will be analyzed by gastrointestinal symptoms questionnaire. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in the gastrointestinal symptoms means better outcome.
Change of gastrointestinal symptoms from baseline to week 12 | The Time Frame contains two time points: Clinical Investigation day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in gastrointestinal symptoms of participants will be analyzed by gastrointestinal symptoms questionnaire. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in the gastrointestinal symptoms means better outcome.
Change of gastrointestinal symptoms from week 4 to week 8 | The Time Frame contains two time points: Clinical Investigation day 2 (after 4 weeks of intervention) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  The change in gastrointestinal symptoms of participants will be analyzed by gastrointestinal symptoms questionnaire. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in the gastrointestinal symptoms means better outcome.
Change of gastrointestinal symptoms from week 8 to week 12 | The Time Frame contains two time points: Clinical Investigation day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  The change in gastrointestinal symptoms of participants will be analyzed by gastrointestinal symptoms questionnaire. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in the gastrointestinal symptoms means better outcome.
Bar acceptance at week 12 | The Time Frame contains Clinical Investigation Day 4 (after 12 weeks of intervention).
  Bar acceptance will be analyzed by acceptance questionnaire.
Change of bar consumption record from baseline to week 4 | The Time Frame contains Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 2 (after 4 weeks of intervention).
  Change of bar consumption will be analyzed by bar consumption record.
Change of bar consumption record from baseline to week 8 | The Time Frame contains Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of bar consumption will be analyzed by bar consumption record.
Change of bar consumption record from baseline to week 12 | The Time Frame contains Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bar consumption will be analyzed by bar consumption record.
Change of bar consumption record from week 4 to week 8 | The Time Frame contains Clinical Investigation Day 2 (after 4 weeks of intervention) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of bar consumption will be analyzed by bar consumption record.
Change of bar consumption record from week 8 to week 12 | The Time Frame contains Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of bar consumption will be analyzed by bar consumption record.
Change in urine and feces hydroxyproline concentration from baseline to week 8 | The Time Frame contains Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 3 (after 8 weeks of intervention).
  Change of hydroxyproline concentration will be analyzed at week 8 by colorimetry technique if significant differences are found in weight loss at week 8
Change in urine and feces hydroxyproline concentration from baseline to week 12 | The Time Frame contains Clinical Investigation Day 1 (at baseline) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of hydroxyproline concentration will be analyzed by colorimetry technique
Change in urine and feces hydroxyproline concentration from week 8 to week 12 | The Time Frame contains Clinical Investigation Day 3 (after 8 weeks of intervention) compared to Clinical Investigation Day 4 (after 12 weeks of intervention).
  Change of hydroxyproline concentration will be analyzed at week 8 by colorimetry technique if significant differences are found in weight loss at week 8

CONTACTS AND LOCATIONS:
Overall Officials: María Ángeles Zulet, Professor, Principal Investigator — Center for Nutrition Research, University of Navarra.; Carlos J González Navarro, PhD, Study Chair — Center for Nutrition Research, University of Navarra.; Fermín I Milagro Yoldi, PhD, Study Chair — Center for Nutrition Research, University of Navarra.; Idoia Ibero Baraibar, PhD, Study Chair — Center for Nutrition Research, University of Navarra.; Itziar Abete Goñi, PhD, Study Chair — Center for Nutrition Research, University of Navarra.; Miguel López Yoldi, PhD, Study Chair — Center for Nutrition Research, University of Navarra.
Locations (1):
- Center for Nutrition Research. University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No